CLINICAL TRIAL: NCT01324570
Title: An Open-label, Multicenter Study of the Safety, Pharmacokinetics, and Efficacy of Buprenorphine Transdermal System (BTDS) in Children From 7 to 16 Years of Age, Inclusive, Who Require Continuous Opioid Analgesia for Moderate to Severe Pain
Brief Title: Safety, Pharmacokinetics (PK), and Efficacy of Buprenorphine Transdermal System (BTDS) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3031; 2010-021954-21 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-29 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Pain
Keywords: Pain; Opioid; Analgesia; Moderate to severe pain
MeSH Terms: conditions — Pain; Agnosia | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overall BTDS (Experimental): Buprenorphine transdermal system
  Interventions: Drug: Buprenorphine transdermal system

INTERVENTIONS:
Drug: Buprenorphine transdermal system — Buprenorphine transdermal system 2.5 mcg/h, 5 mcg/h, 10 mcg/h or 20 mcg/h applied transdermally for 7-day wear.
  Other Names: Butrans

SUMMARY:
The purpose of this study is to characterize the safety, PK, and efficacy of BTDS in patients of ages 7 to 16 years.

DETAILED DESCRIPTION:
A study of safety, PK, and efficacy of BTDS in patients of ages 7 to 16 years, inclusive, who require continuous opioid analgesia for moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female patients, 7 to 16 years of age, inclusive, with malignant and/or nonmalignant moderate to severe pain requiring or anticipated to require continuous, around-the-clock, opioid treatment for at least 2 weeks (based on the investigator's judgment);
* Patients must have written informed consent provided by the parent or legal guardian and assent provided by the patient, when appropriate;
* Patients on incoming opioids must be taking ≤ 80 mg/day morphine or equivalent if aged 12 to 16 years or ≤ 40 mg/day morphine or equivalent if aged 7 to 11 years prior to the screening visit;
* Patients and patient's parent/caregiver must be compliant with the protocol, ie, must be able to perform study assessments and understand and complete the age-appropriate scale to rate pain intensity. Patients must not have a cognitive developmental delay or any other condition that would preclude them from completing the age-appropriate pain scale.

Exclusion Criteria include:

* Patients who are allergic to buprenorphine or have a history of allergies to other opioids (this criterion does not include patients who have experienced common opioid side effects [eg, nausea, constipation]) or who have allergies or other contraindications to transdermal delivery systems or patch adhesives;
* Patients with a dermatological disorder, including burn and skin graft sites, at any relevant patch application site that would preclude proper placement and/or rotation of BTDS patches;
* Patients with evidence of impaired renal function;
* Patients with hepatic impairment;
* Patients with history of seizures;
* Patients with intracranial pressure;
* Patients who have a history of sleep apnea within the past year;
* Patients who require mechanical ventilation during study treatment period, are cyanotic, or who have unstable respiratory disease;
* Patients with clinically significant structural heart disease or a pacemaker;
* Patients with clinically unstable cardiac disease;
* Patients who receive or anticipate to receive investigational medication/therapy during study drug treatment period.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Health Center, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Howard University Hospital, Washington D.C., District of Columbia
  - Jackson Memorial Hospital / University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Kosair Charities Pediatric Clinical Research Unit - University of Louisville, Louisville, Kentucky
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - WCMC, Department of Pediatrics - Hematology/Oncology, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Vidant Medical Center, Greenville, North Carolina
  - The Center for Clinical Research - Carolina Pain Institute, Winston-Salem, North Carolina
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Department of Pediatrics, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Blood and Cancer Center, Austin, Texas
  - Road Runner Research, Ltd., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit: 23-July-2012; Last Patient Last Visit: 23-May-2016. The study was conducted at 33 study centers in the United States
Groups:
- 7 to 11 Years: Children 7 to 11 years of age
- 12 to 16 Years: Children 12 to 16 years of age
Period: Overall Study
Arm/Group | 7 to 11 Years | 12 to 16 Years
Started | 6 | 35
Completed | 2 | 21
Not Completed | 4 | 14
Not completed — Adverse Event | 4 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Confirmed or suspected diversion | 0 | 1
Not completed — Administrative | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population (N=41) was the group of patients who received at least 1 dose of study drug during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 7 to 11 Years | 12 to 16 Years | Total
Number analyzed (Participants) | 6 | 35 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (1.21) | 14.6 (1.31) | 14.0 (1.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 23 | 26
  Male | 3 | 12 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 18 | 21
  Black or African American | 2 | 15 | 17
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety
Description: Safety assessments consisted of reports of AEs, vital signs (blood pressure, pulse rate, respiratory rate, and temperature), weight, hemoglobin-oxygen saturation measured by pulse oximetry (SpO2), clinical laboratory tests, somnolence (assessed by the University of Michigan Sedation Scale [UMSS]), conventional 12-lead electrocardiograms (ECGs), and 24-hour digital 12-lead ECGs (Holter monitor). Safety variables were summarized descriptively within age group for the safety population.
Time Frame: Up to 28 weeks
Population: The safety population (N=41) was the group of patients who received at least 1 dose of study drug during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 7 to 11 Years | 12 to 16 Years
Number analyzed (Participants) | 6 | 35
Participants
  Serious adverse events | 5 | 5
  All other adverse events in ≥ 5% of patients | 6 | 20

2. Primary Outcome: Pharmacokinetics (PK) of Buprenorphine Following Transdermal Administration: Apparent Clearance (CL/F)
Description: The population PK (PopPK) of BTDS buprenorphine in pediatric patients ages 7 to 16 years was described by a 2-compartment model with sequential zero- and first-order absorption from the patch. A fixed allometric relationship was used to describe the effects of changes in ideal body weight (IBW) across pediatric patients on all clearance and volume parameters. Given the sparse sample collections, small sample size, and complexity of the absorption process with the patch formulation, this PopPK model was fit to the pediatric data using nonlinear mixed effects modeling (NONMEM) Bayes method with selective use of priors from previous adult PopPK results. Estimates of fixed effects from the final model were used to calculate the CL/F after patch dosing given the covariate distribution in the PopPK dataset and the typical weights from children in the National Health and Nutrition Examination Survey (NHANES) dataset.
Time Frame: Day 1, end of week 1, days 9/10, end of week 2, and end of week 4 or at discontinuation prior to end of study visit
Population: The full analysis population (FAP) for PK consisted of patients who received study drug and had at least 1 valid quantifiable PK blood sample (N=41).Three patients had no quantifiable plasma buprenorphine concentration measurements and were not included in the PK analysis.The final buprenorphine pediatric PK analysis dataset comprised 38 patients.
Measure: Mean (95% Confidence Interval); unit: Liters/hour
Groups:
- Population PK Analysis Set: Children 7 to 16 years of age (reference patient with IBW of 70 kg)
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 38
Liters/hour | 293 [264 to 326]

3. Secondary Outcome: Pain Right Now Assessment by Patients Aged 7 to 11 Years, Inclusive
Description: Pain right now was assessed using the Faces of Pain Scale-Revised (FPS-R). The FPS-R is a horizontal row of 6 faces representing pain intensity, with "no hurt" at the far left and "hurts worst" at the far right; the intensities are scored as 0, 2, 4, 6, 8, or 10. A score of 0=no pain, and 10=very much pain. For screening to week 4, pain right now was assessed at 30 minutes before initial BTDS application on day 1; one hour after initial BTDS application on day 1; thereafter, once daily at approximately 8 PM for the first 4 weeks. Baseline score was the last assessment prior to the first dose. For weeks 1-4, weekly averages of the pain right now scores were calculated using the sum of all available pain right now scores recorded daily during a given week divided by the number of available scores.
  The study measured pain right now for weeks 6-24 once a week at approximately 8 PM while on treatment; however, no patients in this age group were treated beyond week 12.
Time Frame: Up to 24 weeks
Population: The full analysis population (FAP) was the group of patients who received at least 1 dose of the study drug during the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 7 to 11 Years
Number analyzed (Participants) | 5
units on a scale
  Baseline | 2.80 (1.497)
  Week 1 | 3.49 (1.768)
  Week 2: number analyzed (Participants) | 3
  Week 2 | 2.98 (1.871)
  Week 3: number analyzed (Participants) | 2
  Week 3 | 0.29 (0.000)
  Week 4: number analyzed (Participants) | 2
  Week 4 | 0.00 (0.000)
  Week 5: number analyzed (Participants) | 1
  Week 5 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 6: number analyzed (Participants) | 1
  Week 6 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 7: number analyzed (Participants) | 1
  Week 7 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 8: number analyzed (Participants) | 1
  Week 8 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 9: number analyzed (Participants) | 1
  Week 9 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 10: number analyzed (Participants) | 1
  Week 10 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 11: number analyzed (Participants) | 1
  Week 11 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.
  Week 12: number analyzed (Participants) | 1
  Week 12 | 0.00 (NA) — Since only one patient reported a pain score, standard error was not calculated.

4. Secondary Outcome: Pain Right Now Assessment by Patients Aged 12 to 16 Years, Inclusive
Description: Pain right now was assessed using a 100-mm visual analogue scale (VAS). The 100-mm VAS is a 100-mm line with 1 end marked as "no pain" and the other marked as "pain as bad as it could be." The patient was asked to make a mark on that line indicating his or her level of pain. Pain right now score was defined as the distance (in mm) from the "no pain" end to the patient's mark; 0=no pain and bigger numbers indicate more pain. For screening to week 4, pain right now was assessed 30 minutes before initial BTDS application on day 1; one hour after initial BTDS application on day 1; thereafter, once daily at approximately 8 PM for the first 4 weeks. Baseline was the last assessment prior to the first dose. For weeks 1-4, weekly averages of the pain right now scores were calculated using the sum of all available pain right now scores recorded daily during a given week divided by the number of available scores.
  For weeks 6-24, pain right now was measured once a week at approximately 8 PM.
Time Frame: Up to 24 weeks
Population: The FAP was the group of patients who received at least 1 dose of the study drug during the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 12 to 16 Years
Number analyzed (Participants) | 35
units on a scale
  Baseline: number analyzed (Participants) | 33
  Baseline | 46.6 (4.55)
  Week 1 | 43.1 (4.03)
  Week 2 | 41.6 (4.67)
  Week 3: number analyzed (Participants) | 31
  Week 3 | 36.0 (4.82)
  Week 4: number analyzed (Participants) | 29
  Week 4 | 34.7 (5.09)
  Week 5: number analyzed (Participants) | 23
  Week 5 | 30.3 (5.90)
  Week 6: number analyzed (Participants) | 19
  Week 6 | 28.0 (6.56)
  Week 7: number analyzed (Participants) | 19
  Week 7 | 29.1 (5.56)
  Week 8: number analyzed (Participants) | 16
  Week 8 | 34.3 (7.17)
  Week 9: number analyzed (Participants) | 13
  Week 9 | 27.3 (5.83)
  Week 10: number analyzed (Participants) | 17
  Week 10 | 36.7 (5.83)
  Week 11: number analyzed (Participants) | 14
  Week 11 | 35.7 (8.15)
  Week 12: number analyzed (Participants) | 15
  Week 12 | 42.5 (8.31)
  Week 13: number analyzed (Participants) | 15
  Week 13 | 36.0 (7.99)
  Week 14: number analyzed (Participants) | 13
  Week 14 | 38.2 (8.67)
  Week 15: number analyzed (Participants) | 12
  Week 15 | 30.5 (6.52)
  Week 16: number analyzed (Participants) | 12
  Week 16 | 38.7 (6.94)
  Week 17: number analyzed (Participants) | 14
  Week 17 | 30.9 (5.74)
  Week 18: number analyzed (Participants) | 15
  Week 18 | 37.7 (6.88)
  Week 19: number analyzed (Participants) | 14
  Week 19 | 37.4 (5.50)
  Week 20: number analyzed (Participants) | 12
  Week 20 | 35.6 (7.48)
  Week 21: number analyzed (Participants) | 16
  Week 21 | 32.4 (5.97)
  Week 22: number analyzed (Participants) | 16
  Week 22 | 38.1 (5.84)
  Week 23: number analyzed (Participants) | 15
  Week 23 | 38.7 (6.42)
  Week 24: number analyzed (Participants) | 11
  Week 24 | 36.5 (5.35)

5. Secondary Outcome: Parent/Caregiver-assessed Global Impression of Change (PGIC)
Description: The PGIC rating score variable was collected on a 7-point scale ranging from 1 to 7 (where 1 = very much improved; and 7 = very much worse). The PGIC is designed to assess overall satisfaction with the treatment. The PGIC score was summarized using the number and percent of patients in each of the 7 possible response categories overall and by age group. PGIC was assessed by the parent/caregiver at the end of treatment visit or early discontinuation visit.
Time Frame: End of treatment (week 24) or early discontinuation visit
Population: The full analysis population (FAP) (N=40) was the group of patients who received at least 1 dose of the study drug during the study; however data was provided for only 38 patients for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 7 to 11 Years | 12 to 16 Years
Number analyzed (Participants) | 4 | 34
Participants
  Participants Represented | 4 | 34
  1 = Very much improved | 1 | 6
  2 = Much improved | 0 | 12
  3 = Minimally improved | 0 | 8
  4 = No change | 2 | 5
  5 = Minimally worse | 1 | 2
  6 = Much worse | 0 | 1
  7 = Very much worse | 0 | 0

6. Primary Outcome: Pharmacokinetics (PK) of Buprenorphine Following Transdermal Administration: Apparent Volume of Distribution (Vc/F)
Description: The population PK (PopPK) of BTDS buprenorphine in pediatric patients ages 7 to 16 years was described by a 2-compartment model with sequential zero- and first-order absorption from the patch. A fixed allometric relationship was used to describe the effects of changes in ideal body weight (IBW) across pediatric patients on all clearance and volume parameters. Given the sparse sample collections, small sample size, and complexity of the absorption process with the patch formulation, this PopPK model was fit to the pediatric data using nonlinear mixed effects modeling (NONMEM) Bayes method with selective use of priors from previous adult PopPK results. Estimates of fixed effects from the final model were used to calculate the Vc/F after patch dosing given the covariate distribution in the PopPK dataset and the typical weights from children in the National Health and Nutrition Examination Survey (NHANES) dataset.
Time Frame: Day 1, end of week 1, days 9/10, end of week 2, and end of week 4 or at discontinuation prior to end of study visit
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 38
Liters | 2350 [1950 to 2820]

ADVERSE EVENTS:
Time Frame: Non-serious treatment-emergent adverse events (TEAEs) were collected from the initiation of treatment with study drug up to 7 days after the last dose of study drug. Serious adverse events (SAEs) were collected from the signing of the informed consent form through 30 days of the last dose of study drug.
Description: For the assessment of SAEs and TEAEs, the analysis population included all patients exposed to at least 1 dose of study drug (ie, safety population).
  An SAE of pneumohemothorax occurred in 1 patient during screening and an SAE of sickle cell pain crisis occurred in 1 patient during screening. Both patients were considered screen failures, were not treated with study drug, and were not included in the safety population.
Arm/Group | 7 to 11 Years | 12 to 16 Years
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/35
Serious Adverse Events (participants affected / at risk) | 5/6 | 5/35
Other Adverse Events (participants affected / at risk) | 6/6 | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 7 to 11 Years (N=6) | 12 to 16 Years (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Hereditary Angioedema (Congenital, familial and genetic disorders) | 0 | 1
Sickle Cell Anaemia With Crisis (Congenital, familial and genetic disorders) | 0 | 2
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Osteomyelitis Chronic (Infections and infestations) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 7 to 11 Years (N=6) | 12 to 16 Years (N=35)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 7
Application Site Pruritus (General disorders) | 0 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Application Site Irritation (General disorders) | 1 | 4
Fatigue (General disorders) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 5
Dizziness (Nervous system disorders) | 1 | 2
Paresthesia (Nervous system disorders) | 0 | 2
Sedation (Nervous system disorders) | 1 | 0
Sickle Cell Anaemia With Crisis (Congenital, familial and genetic disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Patient recruitment in the younger age group was difficult and the sample size is smaller than the older age group. This limitation should be a consideration when interpreting the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days